CLINICAL TRIAL: NCT00544570
Title: High Dose Sequential Therapy for Poor Risk Recurrent or Refractory Hodgkin's Disease
Brief Title: High-Dose Chemotherapy in Treating Patients Undergoing Stem Cell Transplant for Recurrent or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Eileen Smith MD, City of Hope Medical Center
Purpose: Treatment
Other Study IDs: CDR0000567466; P30CA033572 (NIH); P01CA030206 (NIH); CHNMC-97160
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Filgrastim; Carmustine; Cyclophosphamide; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy; Whole-Body Irradiation

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cyclophosphamide
Drug: etoposide
Drug: melphalan
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving high-dose chemotherapy before a peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or by killing them. Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected and stored. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by high-dose chemotherapy and radiation therapy.

PURPOSE: This clinical trial is studying the side effects and how well high-dose chemotherapy works in treating patients undergoing stem cell transplant for recurrent or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the feasibility and toxicity of high-dose sequential therapy comprising high-dose etoposide and cyclophosphamide with filgrastim (G-CSF) support followed by 2 courses of high-dose therapy and autologous stem cell transplantation in patients with poor-risk recurrent or refractory Hodgkin lymphoma.
* To analyze the response rate, progression-free survival, and overall survival of patients treated with this regimen.
* To determine the percentage of patients who can achieve a minimal disease status after two courses of Hodgkin lymphoma chemotherapy and before "classical autologous stem cell transplantation."

OUTLINE:

* First high-dose chemotherapy*: Patients receive high-dose cyclophosphamide IV over 2 hours followed by etoposide IV over 4 hours.

NOTE: *Patients with minimal disease (i.e., a single lymph node ≤ 2 cm in maximal horizontal diameter or a > 75% reduction in a bulky (≥ 10 cm) tumor mass AND no morphological evidence of active bone marrow disease) at initial evaluation do not receive the first high-dose chemotherapy but proceed directly to peripheral blood stem cell (PBSC) mobilization with filgrastim (G-CSF) for 3 days and PBSC collection beginning on day 4.

* Peripheral stem cell mobilization and collection: Patients receive G-CSF subcutaneously beginning 96 hours after completion of etoposide and continuing through completion of PBSC collection. Patients undergo leukapheresis to collect PBSC for reinfusion after additional high-dose therapy.
* Second high-dose chemotherapy: Patients receive high-dose melphalan IV over 30 minutes on day -1.
* First PBSC infusion: At least 24 hours after completion of melphalan, patients undergo reinfusion of PBSC on day 0.
* Local radiotherapy: Patients with a localized tumor mass > 5 cm after the second course of chemotherapy or a previous history of bulky disease (> 10 cm or mediastinal mass > 1/3 of transverse thoracic diameter) that has not been irradiated may receive local radiotherapy for 2 weeks, at the discretion of the principal investigator.
* High-dose therapy: Eight to 12 weeks after completion of the second course of chemotherapy, patients receive 1 of 2 regimens.

  * Regimen A: Patients undergo fractionated total body irradiation 3 times daily on days -8 to -5 (10 fractions) and receive high-dose etoposide IV over 4 hours on day -4 and cyclophosphamide IV on day -2.
  * Regimen B: Patients receive high-dose carmustine IV over 4 hours on days -7 to -5 and etoposide and cyclophosphamide as in regimen A.
* Second PBSC infusion: At least 48 hours after completion of cyclophosphamide, patients undergo reinfusion of PBSC on day 0.

After completion of study therapy, patients are followed at day 60 and then every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin lymphoma

  * Diagnosis reviewed by the participating institution
* Failed to achieve complete remission (CR) after first-line chemotherapy or chemoradiotherapy (i.e., induction failure) OR not felt to be curable by radiotherapy alone
* Relapsed after standard chemotherapy regimen for Hodgkin lymphoma AND has ≥ 1 of the following poor-risk features:

  * Extranodal disease at relapse
  * Interval from first CR to relapse < 12 months
  * B symptoms at relapse
  * Chemo-resistant relapse OR failure to achieve a second CR with conventional nontransplantation salvage chemotherapy regimen
* No cytogenetic abnormality on cytogenetic analysis of bone marrow

PATIENT CHARACTERISTICS:

Inclusion criteria:

* SWOG performance status 0-1
* LVEF > 50% by 2D-ECHO or MUGA scan

  * Patients with LVEF between 45-50% and without wall motion abnormalities are assessed on an individual basis after consultation with the cardiologist
* FEV_1 or DLCO > 45% predicted
* Creatinine clearance > 60 mL/min
* HIV-negative
* Hepatitis B surface antigen-negative
* Hepatitis C virus-negative
* ALT ≤ 5 times upper limit of normal
* No inadequate vital organ function
* No active infection
* Fertile patients must use adequate contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent, post-transplantation, consolidative radiotherapy to residual masses allowed provided the patient has engrafted with a WBC > 4,000/μL and a platelet count > 100,000/μL

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Feasibility
Toxicity as assessed by NCI CTC v2.0

SECONDARY OUTCOMES:
Response rate
Progression-free survival
Overall survival
Percentage of patients who achieve minimal disease status after 2 courses

CONTACTS AND LOCATIONS:
Overall Officials: Eileen P. Smith, MD, Study Chair — City of Hope Comprehensive Cancer Center